CLINICAL TRIAL: NCT04349631
Title: A Phase II, Open Label, Single-Center, Clinical Trial to Assess Safety and Efficacy of HB-adMSCs to Provide Immune Support Against Coronavirus Disease
Brief Title: A Clinical Trial to Determine the Safety and Efficacy of HB-adMSCs to Provide Protection Against COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hope Biosciences Research Foundation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HBCOVID01
Record Dates: First submitted 2020-04-06; First posted 2020-04-16 (Actual); Results first posted 2023-10-31 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: COVID-19
Keywords: Coronavirus; Prevention; Immune support; stem cells; mesenchymal stem cells; adipose-derived mesenchymal stem cells
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HB-adMSCs (Experimental): Five IV infusions of autologous, adipose-derived mesenchymal stem cells. Baseline laboratory data will be collected prior to first infusion; follow-up data will be compared against baseline according to the following schedule: safety lab follow ups at weeks 6, 14, 26; inflammatory marker follow ups at weeks 6, 14, 26; SF-36 and PHQ-9 Questionnaires at weeks 2, 6, 10, 14, 18, 22, 26.
  Interventions: Biological: HB-adMSCs

INTERVENTIONS:
Biological: HB-adMSCs — Five IV infusions of autologous adipose-derived mesenchymal stem cells. Baseline laboratory values will be collected prior to first infusion and compared at following visits. Safety labs will be assessed at weeks 6, 14, 26. Inflammatory markers will be assessed at weeks 6, 14, 26. SF-36 and PHQ-9 questionnaires will be assessed at weeks 2, 6, 10, 14, 18, 22, 26.

SUMMARY:
Hope Biosciences is conducting a research study of an investigational product called autologous adipose-derived mesenchymal stem cells (abbreviated as HB-adMSCs) to provide immune support against COVID-19. The study purpose is to evaluate the safety and efficacy of five IV infusions of HB-adMSCs in subjects with no signs of COVID-19.

DETAILED DESCRIPTION:
This is a Phase II, Open Label, Single-Center, Clinical Trial to Assess Efficacy of HB-adMSCs to Provide Immune Support Against Coronavirus Disease. 51 patients were enrolled. All patients have previously banked their own mesenchymal stem cells at Hope Biosciences. Eligible participants are either 65 years of age or older, have preexisting conditions, or are at high exposure risk of contracting COVID-19. The primary objective of this study is to provide immune support against COVID-19, measured by the presence or absence of adverse events and serious adverse events related to the study drug. In addition, participants will be monitored for overall clinical status by standard clinical laboratories and inflammatory markers. Participants will complete Short Form Health Survey (SF-36) and depression module (PHQ-9) questionnaires.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet the criteria for 1,2, OR 3, AND 4-7 to be eligible.

1. Men, and women 65 years of age or older (according to CDC provisions) OR
2. Participant works in healthcare facility or other well characterized high-risk environment OR
3. Has underlying conditions including but not limited to cardiopathies, diabetes mellitus, cancer, COPD, asthma or any other systemic autoimmune disease.
4. Subject must have previously banked their cells at Hope Biosciences
5. No signs or symptoms of infection, including but not limited to, body temperature >100 F and pulse rate > 100 BPM.
6. Subject provides written informed consent prior to initiation of any study procedures.
7. Agrees to the collection of venous blood per protocol.
8. Agrees to conformational testing for SARS-CoV-2 before end of study.

Exclusion Criteria:

Subjects must not have any of the following criteria to be eligible.

1. Women who are pregnant or lactating, or those who are not pregnant but do not take effective contraceptive measures
2. Patients who are participating in other clinical trials or have intake of investigational drug within the previous 30 days;
3. Inability to provide informed consent or to comply with test requirements;
4. Any medical disease or condition that, in the opinion of the site PI or sub-investigator, precludes study participation. Including acute, subacute, intermittent or chronic medical disease or condition that would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the subject's successful completion of this trial.
5. Patients who have received a stem cell treatment within one year.
6. Receipt of any other SARS-CoV-2 or other experimental coronavirus vaccine at any time prior to or during the study.
7. Patient currently or recently symptomatic for COVID-19 or anyone with COVID-19 associated symptoms within the past 30-days

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2020-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thanh Cheng, MD, Principal Investigator — Hope Biosciences Stem Cell Research Foundation
Locations (1):
- Hope Biosciences Stem Cell Research Foundation, Sugar Land, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HB-adMSCs
Started | 51
Completed | 41
Not Completed | 10
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 7

BASELINE CHARACTERISTICS:
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (18.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 48
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 20
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 31
  More than one race | 0
  Unknown or Not Reported | 0
Age, Customized [Count of Participants; unit: Participants]
  18-60 years | 30
  61-80 years | 18
  > 80 years | 3
Height [Mean (Standard Deviation); unit: centimeters] | 167.59 (9.642)
Weight [Mean (Standard Deviation); unit: kilograms] | 73.05 (17.086)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Hospitalization for COVID-19
Description: Number of subjects that require hospitalization for COVID-19
Time Frame: Week 0 through Week 26 (End of Study)
Population: There was no incidence of hospitalization for COVID-19 in this study. Therefore, the analyses for this outcome measure were not performed.
Measure: Count of Participants; unit: Participants
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 51
Participants | 0

2. Primary Outcome: Incidence of Symptoms for COVID-19
Description: Number of subjects that develop symptoms associated with COVID-19, such as fever, shortness of breath/difficulty breathing, cough
Time Frame: Week 0 through Week 26 (End of Study)
Population: There was no incidence of symptoms for COVID-19 in this study. Therefore, the analyses for this outcome measure were not performed.
Measure: Count of Participants; unit: Participants
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 51
Participants | 0

3. Secondary Outcome: Absence of Upper/Lower Respiratory Infection
Description: Absence of upper/lower respiratory infection (with hospitalization criteria)
Time Frame: Week 0 through Week 26 (End of Study)
Population: There was no upper/lower respiratory infection due to COVID-19 reported in this study. Therefore, the analyses for this outcome measure were not performed.
Measure: Count of Participants; unit: Participants
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 51
Participants | 0

4. Secondary Outcome: Change From Baseline in Glucose
Description: Change from baseline in level of glucose in the blood (mg/dL)
Time Frame: Weeks 0, 6, 14, 26
Population: At baseline (Week 0), the maximum number analyzed was 50. This was the largest N collected.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 50
mg/dL
  Week 0 | 96.4 (16.11)
  Week 6: number analyzed (Participants) | 47
  Week 6 | -4.1 (18.00)
  Week 14: number analyzed (Participants) | 42
  Week 14 | 5.8 (21.07)
  Week 26: number analyzed (Participants) | 40
  Week 26 | 6.8 (40.90)

5. Secondary Outcome: Change From Baseline in Calcium
Description: Change from baseline in level of calcium in the blood (mg/dL)
Time Frame: Weeks 0, 6, 14, 26
Population: At baseline (Week 0), the maximum number analyzed was 51. This was the largest N collected.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 51
mg/dL
  Week 0 | 9.44 (0.410)
  Week 6: number analyzed (Participants) | 47
  Week 6 | -0.03 (0.455)
  Week 14: number analyzed (Participants) | 42
  Week 14 | 0.00 (0.441)
  Week 26: number analyzed (Participants) | 40
  Week 26 | -0.03 (0.394)

6. Secondary Outcome: Change From Baseline in Albumin
Description: Change from baseline in level of albumin in the blood (g/dL)
Time Frame: Weeks 0, 6, 14, 26
Population: At baseline (Week 0), the maximum number analyzed was 51. This was the largest N collected.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 51
g/dL
  Week 0 | 4.62 (0.306)
  Week 6: number analyzed (Participants) | 47
  Week 6 | -0.10 (0.280)
  Week 14: number analyzed (Participants) | 42
  Week 14 | -0.22 (0.301)
  Week 26: number analyzed (Participants) | 40
  Week 26 | -0.05 (0.283)

7. Secondary Outcome: Change From Baseline in Total Protein
Description: Change from baseline in level of total protein in the blood (g/dL)
Time Frame: Weeks 0, 6, 14, 26
Population: At baseline (Week 0), the maximum number analyzed was 51. This was the largest N collected.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 51
g/dL
  Week 0 | 6.89 (0.469)
  Week 6: number analyzed (Participants) | 47
  Week 6 | -0.04 (0.394)
  Week 14: number analyzed (Participants) | 42
  Week 14 | -0.11 (0.500)
  Week 26: number analyzed (Participants) | 40
  Week 26 | 0.02 (0.428)

8. Secondary Outcome: Change From Baseline in Sodium
Description: Change from baseline in level of sodium in the blood (mmol/L)
Time Frame: Weeks 0, 6, 14, 26
Population: At baseline (Week 0), the maximum number analyzed was 51. This was the largest N collected.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 51
mmol/L
  Week 0 | 141.0 (2.11)
  Week 6: number analyzed (Participants) | 47
  Week 6 | -0.7 (2.53)
  Week 14: number analyzed (Participants) | 42
  Week 14 | -1.3 (2.17)
  Week 26: number analyzed (Participants) | 40
  Week 26 | -1.4 (2.29)

9. Secondary Outcome: Change From Baseline in Total Carbon Dioxide
Description: Change from baseline in level of carbon dioxide in the blood (mmol/L)
Time Frame: Weeks 0, 6, 14, 26
Population: At baseline (Week 0), the maximum number analyzed was 51. This was the largest N collected.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 51
mmol/L
  Week 0 | 23.4 (2.80)
  Week 6: number analyzed (Participants) | 47
  Week 6 | 0.9 (2.76)
  Week 14: number analyzed (Participants) | 42
  Week 14 | 0.6 (2.68)
  Week 26: number analyzed (Participants) | 40
  Week 26 | 0.1 (2.92)

10. Secondary Outcome: Change From Baseline in Potassium
Description: Change from baseline in level of potassium in the blood (mmol/L)
Time Frame: Weeks 0, 6, 14, 26
Population: At baseline (Week 0), the maximum number analyzed was 51. This was the largest N collected.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 51
mmol/L
  Week 0 | 4.31 (0.364)
  Week 6: number analyzed (Participants) | 47
  Week 6 | -0.21 (0.409)
  Week 14: number analyzed (Participants) | 42
  Week 14 | -0.16 (0.369)
  Week 26: number analyzed (Participants) | 40
  Week 26 | -0.10 (0.415)

11. Secondary Outcome: Change From Baseline in Chloride
Description: Change from baseline in level of chloride in the blood (mmol/L)
Time Frame: Weeks 0, 6, 14, 26
Population: At baseline (Week 0), the maximum number analyzed was 51. This was the largest N collected.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 51
mmol/L
  Week 0 | 102.0 (2.73)
  Week 6: number analyzed (Participants) | 47
  Week 6 | -0.7 (2.82)
  Week 14: number analyzed (Participants) | 42
  Week 14 | 0.1 (2.39)
  Week 26: number analyzed (Participants) | 40
  Week 26 | -0.4 (2.37)

12. Secondary Outcome: Change From Baseline in Blood Urea Nitrogen (BUN)
Description: Change from baseline in level of blood urea nitrogen (BUN) in the blood (mg/dL)
Time Frame: Weeks 0, 6, 14, 26
Population: At baseline (Week 0), the maximum number analyzed was 51. This was the largest N collected.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 51
mg/dL
  Week 0 | 15.0 (4.21)
  Week 6: number analyzed (Participants) | 47
  Week 6 | -1.0 (3.22)
  Week 14: number analyzed (Participants) | 42
  Week 14 | 0.5 (3.67)
  Week 26: number analyzed (Participants) | 40
  Week 26 | -0.7 (3.61)

13. Secondary Outcome: Change From Baseline in Creatinine
Description: Change from baseline in level of creatinine in the blood (mg/dL)
Time Frame: Weeks 0, 6, 14, 26
Population: At baseline (Week 0), the maximum number analyzed was 51. This was the largest N collected.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 51
mg/dL
  Week 0 | 0.838 (0.1946)
  Week 6: number analyzed (Participants) | 47
  Week 6 | -0.003 (0.1007)
  Week 14: number analyzed (Participants) | 42
  Week 14 | -0.000 (0.1383)
  Week 26: number analyzed (Participants) | 40
  Week 26 | -0.013 (0.0895)

14. Secondary Outcome: Change From Baseline in Alkaline Phosphatase
Description: Change from baseline in level of alkaline phosphatase in the blood (IU/L)
Time Frame: Weeks 0, 6, 14, 26
Population: At baseline (Week 0), the maximum number analyzed was 51. This was the largest N collected.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 51
IU/L
  Week 0 | 61.9 (20.56)
  Week 6: number analyzed (Participants) | 47
  Week 6 | -1.0 (6.69)
  Week 14: number analyzed (Participants) | 42
  Week 14 | -2.3 (6.50)
  Week 26: number analyzed (Participants) | 40
  Week 26 | 5.3 (9.59)

15. Secondary Outcome: Change From Baseline in Alanine Aminotransferase
Description: Change from baseline in level of alanine aminotransferase in the blood (IU/L)
Time Frame: Weeks 0, 6, 14, 26
Population: At baseline (Week 0), the maximum number analyzed was 51. This was the largest N collected.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 51
IU/L
  Week 0 | 21.2 (8.87)
  Week 6: number analyzed (Participants) | 47
  Week 6 | -2.0 (4.95)
  Week 14: number analyzed (Participants) | 42
  Week 14 | -3.2 (5.55)
  Week 26: number analyzed (Participants) | 40
  Week 26 | -1.1 (6.82)

16. Secondary Outcome: Change From Baseline in Aspartate Aminotransferase
Description: Change from baseline in level of aspartate aminotransferase in the blood (IU/L)
Time Frame: Weeks 0, 6, 14, 26
Population: At baseline (Week 0), the maximum number analyzed was 51. This was the largest N collected.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 51
IU/L
  Week 0 | 22.7 (6.77)
  Week 6: number analyzed (Participants) | 47
  Week 6 | -3.3 (6.37)
  Week 14: number analyzed (Participants) | 42
  Week 14 | -3.1 (6.26)
  Week 26: number analyzed (Participants) | 40
  Week 26 | -0.1 (6.03)

17. Secondary Outcome: Change From Baseline in Total Bilirubin
Description: Change from baseline in level of total bilirubin in the blood (mg/dL)
Time Frame: Weeks 0, 6, 14, 26
Population: At baseline (Week 0), the maximum number analyzed was 51. This was the largest N collected.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 51
mg/dL
  Week 0 | 0.50 (0.338)
  Week 6: number analyzed (Participants) | 41
  Week 6 | -0.03 (0.185)
  Week 14: number analyzed (Participants) | 36
  Week 14 | -0.03 (0.212)
  Week 26: number analyzed (Participants) | 33
  Week 26 | -0.05 (0.195)

18. Secondary Outcome: Change From Baseline in Leukocytes
Description: Change from baseline in level of leukocytes in the blood (x 10^9/L)
Time Frame: Weeks 0, 6, 14, 26
Population: At baseline (Week 0), the maximum number analyzed was 51. This was the largest N collected.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 51
10^9 cells/L
  Week 0 | 6.41 (1.888)
  Week 6: number analyzed (Participants) | 48
  Week 6 | -0.13 (1.397)
  Week 14: number analyzed (Participants) | 42
  Week 14 | 0.07 (1.248)
  Week 26: number analyzed (Participants) | 40
  Week 26 | 0.01 (1.553)

19. Secondary Outcome: Change From Baseline in Erythrocytes
Description: Change from baseline in erythrocytes in the blood (10^12/L)
Time Frame: Weeks 0, 6, 14, 26
Population: At baseline (Week 0), the maximum number analyzed was 51. This was the largest N collected.
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 51
10^12 cells/L
  Week 0 | 4.610 (0.5315)
  Week 6: number analyzed (Participants) | 48
  Week 6 | 0.018 (0.2687)
  Week 14: number analyzed (Participants) | 42
  Week 14 | -0.015 (0.2871)
  Week 26: number analyzed (Participants) | 40
  Week 26 | 0.042 (0.2340)

20. Secondary Outcome: Change From Baseline in Hemoglobin
Description: Change from baseline in level of hemoglobin in the blood (g/dL)
Time Frame: Weeks 0, 6, 14, 26
Population: At baseline (Week 0), the maximum number analyzed was 51. This was the largest N collected.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 51
g/dL
  Week 0 | 13.83 (1.702)
  Week 6: number analyzed (Participants) | 48
  Week 6 | -0.02 (0.789)
  Week 14 | -0.22 (0.931)
  Week 26 | 0.03 (0.814)

21. Secondary Outcome: Change From Baseline in Hematocrit
Description: Change from baseline in level of hematocrit in the blood (%)
Time Frame: Weeks 0, 6, 14, 26
Population: At baseline (Week 0), the maximum number analyzed was 51. This was the largest N collected.
Measure: Mean (Standard Deviation); unit: percentage of erythrocytes
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 51
percentage of erythrocytes
  Week 0 | 43.27 (4.636)
  Week 6 | -0.70 (2.757)
  Week 14 | -1.60 (2.991)
  Week 26 | -1.06 (2.737)

22. Secondary Outcome: Change From Baseline in Mean Corpuscular Volume
Description: Change from baseline in mean corpuscular volume in the blood (fL)
Time Frame: Weeks 0, 6, 14, 26
Population: At baseline (Week 0), the maximum number analyzed was 51. This was the largest N collected.
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 51
fL
  Week 0 | 94.2 (6.35)
  Week 6 | -2.0 (2.81)
  Week 14 | -3.1 (3.86)
  Week 26 | -3.2 (3.82)

23. Secondary Outcome: Change From Baseline in Mean Corpuscular Hemoglobin
Description: Change from baseline in mean corpuscular hemoglobin in the blood (pg)
Time Frame: Weeks 0, 6, 14, 26
Population: At baseline (Week 0), the maximum number analyzed was 51. This was the largest N collected.
Measure: Mean (Standard Deviation); unit: pg
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 51
pg
  Week 0 | 30.05 (2.119)
  Week 6: number analyzed (Participants) | 48
  Week 6 | -0.15 (0.697)
  Week 14: number analyzed (Participants) | 42
  Week 14 | -0.33 (0.530)
  Week 26: number analyzed (Participants) | 40
  Week 26 | -0.17 (1.004)

24. Secondary Outcome: Change From Baseline in Mean Corpuscular Hemoglobin Concentration
Description: Change from baseline in mean corpuscular hemoglobin in the blood (g/dL)
Time Frame: Weeks 0, 6, 14, 26
Population: At baseline (Week 0), the maximum number analyzed was 51. This was the largest N collected.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 51
g/dL
  Week 0 | 31.94 (1.401)
  Week 6: number analyzed (Participants) | 48
  Week 6 | 0.47 (1.097)
  Week 14: number analyzed (Participants) | 42
  Week 14 | 0.70 (1.476)
  Week 26: number analyzed (Participants) | 40
  Week 26 | 0.88 (1.292)

25. Secondary Outcome: Change From Baseline in Erythrocyte Distribution Width
Description: Change from baseline in erythrocyte distribution width in the blood (%)
Time Frame: Weeks 0, 6, 14, 26
Population: At baseline (Week 0), the maximum number analyzed was 51. This was the largest N collected.
Measure: Mean (Standard Deviation); unit: % of erythrocytes
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 51
% of erythrocytes
  Week 0 | 14.00 (1.739)
  Week 6: number analyzed (Participants) | 48
  Week 6 | -1.09 (1.628)
  Week 14: number analyzed (Participants) | 42
  Week 14 | -1.14 (0.965)
  Week 26: number analyzed (Participants) | 40
  Week 26 | -1.00 (0.804)

26. Secondary Outcome: Change From Baseline in Neutrophils
Description: Change from baseline in neutrophils in the blood (%) (leukocyte differential)
Time Frame: Weeks 0, 6, 14, 26
Population: At baseline (Week 0), the maximum number analyzed was 44. This was the largest N collected.
Measure: Mean (Standard Deviation); unit: percentage of neutrophils in the blood
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 44
percentage of neutrophils in the blood
  Week 0 | 59.2 (8.62)
  Week 6 | -0.70 (8.123)
  Week 14: number analyzed (Participants) | 42
  Week 14 | -0.40 (8.121)
  Week 26: number analyzed (Participants) | 40
  Week 26 | -1.10 (8.111)

27. Secondary Outcome: Change From Baseline in Lymphocytes
Description: Change from baseline in lymphocytes in the blood (%) (leukocyte differential)
Time Frame: Weeks 0, 6, 14, 26
Population: At baseline (Week 0), the maximum number analyzed was 44. This was the largest N collected.
Measure: Mean (Standard Deviation); unit: percentage of lymphocytes in the blood
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 44
percentage of lymphocytes in the blood
  Week 0 | 30.5 (8.15)
  Week 6 | 0.27 (7.049)
  Week 14: number analyzed (Participants) | 42
  Week 14 | -0.19 (7.487)
  Week 26: number analyzed (Participants) | 40
  Week 26 | 0.63 (7.413)

28. Secondary Outcome: Change From Baseline in Monocytes
Description: Change from baseline in monocytes in the blood (%) (leukocyte differential)
Time Frame: Weeks 0, 6, 14, 26
Population: At baseline (Week 0), the maximum number analyzed was 44. This was the largest N collected.
Measure: Mean (Standard Deviation); unit: percentage of monocytes in the blood
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 44
percentage of monocytes in the blood
  Week 0 | 7.3 (1.85)
  Week 6 | 0.05 (1.765)
  Week 14: number analyzed (Participants) | 42
  Week 14 | 0.29 (1.384)
  Week 26: number analyzed (Participants) | 40
  Week 26 | 0.03 (1.387)

29. Secondary Outcome: Change From Baseline in Eosinophils
Description: Change from baseline in eosinophils in the blood (%) (leukocyte differential)
Time Frame: Weeks 0, 6, 14, 26
Population: At baseline (Week 0), the maximum number analyzed was 44. This was the largest N collected.
Measure: Mean (Standard Deviation); unit: percentage of eosinophils in the blood
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 44
percentage of eosinophils in the blood
  Week 0 | 2.3 (2.14)
  Week 6 | 0.23 (1.118)
  Week 14: number analyzed (Participants) | 42
  Week 14 | -0.02 (1.440)
  Week 26: number analyzed (Participants) | 40
  Week 26 | -0.03 (1.577)

30. Secondary Outcome: Change From Baseline in Basophils
Description: Change from baseline in basophils in the blood (%) (leukocyte differential)
Time Frame: Weeks 0, 6, 14, 26
Population: At baseline (Week 0), the maximum number analyzed was 44. This was the largest N collected.
Measure: Mean (Standard Deviation); unit: percentage of basophils in the blood
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 44
percentage of basophils in the blood
  Week 0 | 0.6 (0.55)
  Week 6 | 0.18 (0.540)
  Week 14: number analyzed (Participants) | 42
  Week 14 | 0.29 (0.457)
  Week 26: number analyzed (Participants) | 40
  Week 26 | 0.25 (0.439)

31. Secondary Outcome: Change From Baseline in Platelets
Description: Change from baseline in platelets in the blood (x 10^9/L)
Time Frame: Weeks 0, 6, 14, 26
Population: At baseline (Week 0), the maximum number analyzed was 51. This was the largest N collected.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 51
10^9 cells/L
  Week 0 | 268.8 (73.48)
  Week 6: number analyzed (Participants) | 48
  Week 6 | -0.3 (30.85)
  Week 14: number analyzed (Participants) | 42
  Week 14 | -1.9 (29.50)
  Week 26: number analyzed (Participants) | 40
  Week 26 | -11.6 (26.06)

32. Secondary Outcome: Change From Baseline in Prothrombin Time
Description: Change from baseline in prothrombin time in the blood (seconds)
Time Frame: Weeks 0, 6, 14, 26
Population: At baseline (Week 0), the maximum number analyzed was 47. This was the largest N collected.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 47
seconds
  Week 0 | 11.16 (0.663)
  Week 6: number analyzed (Participants) | 43
  Week 6 | -0.08 (0.596)
  Week 14: number analyzed (Participants) | 40
  Week 14 | 0.20 (0.647)
  Week 26: number analyzed (Participants) | 38
  Week 26 | 0.49 (0.766)

33. Secondary Outcome: Change From Baseline in International Normalized Ratio (INR)
Description: Change from baseline in international normalized ratio in the blood (INR) (ratio)
Time Frame: Weeks 0, 6, 14, 26
Population: At baseline (Week 0), the maximum number analyzed was 47. This was the largest N collected.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 47
ratio
  Week 0 | 1.06 (0.077)
  Week 6: number analyzed (Participants) | 43
  Week 6 | -0.01 (0.074)
  Week 14: number analyzed (Participants) | 40
  Week 14 | 0.03 (0.078)
  Week 26: number analyzed (Participants) | 38
  Week 26 | 0.08 (0.093)

34. Secondary Outcome: Change From Baseline in Tumor Necrosis Factor Alpha (TNF-alpha)
Description: Change from baseline in tumor necrosis factor alpha (TNF-alpha) in the blood (ng/L)
Time Frame: Weeks 0, 6, 14, 26
Population: At baseline (Week 0), the maximum number analyzed was 44. This was the largest N collected.
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 44
ng/L
  Week 0 | 1.75 (4.974)
  Week 6: number analyzed (Participants) | 43
  Week 6 | 0.02 (0.902)
  Week 14: number analyzed (Participants) | 40
  Week 14 | -0.12 (0.759)
  Week 26: number analyzed (Participants) | 39
  Week 26 | -0.26 (1.271)

35. Secondary Outcome: Change From Baseline in Interleukin-6
Description: Change from baseline in Interleukin-6 in the blood (ng/L)
Time Frame: Weeks 0, 6, 14, 26
Population: At baseline (Week 0), the maximum number analyzed was 33. This was the largest N collected.
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 33
ng/L
  Week 0 | 2.5 (2.07)
  Week 6: number analyzed (Participants) | 31
  Week 6 | 0.78 (3.071)
  Week 14: number analyzed (Participants) | 29
  Week 14 | 0.59 (2.938)
  Week 26: number analyzed (Participants) | 24
  Week 26 | -0.50 (2.344)

36. Secondary Outcome: Change From Baseline in Interleukin-10
Description: Change from baseline in Interleukin-10 in the blood (ng/L)
Time Frame: Weeks 0, 6, 14, 26
Population: At baseline (Week 0), the maximum number analyzed was 27. This was the largest N collected.
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 27
ng/L
  Week 0 | 6.1 (2.62)
  Week 6: number analyzed (Participants) | 15
  Week 6 | 1.63 (2.483)
  Week 14: number analyzed (Participants) | 19
  Week 14 | 0.83 (3.074)
  Week 26: number analyzed (Participants) | 14
  Week 26 | 7.99 (21.579)

37. Secondary Outcome: Change From Baseline in C-Reactive Protein
Description: Change from baseline in C-Reactive Protein in the blood (mg/dL)
Time Frame: Weeks 0, 6, 14, 26
Population: At baseline (Week 0), the maximum number analyzed was 24. This was the largest N collected.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 24
mg/dL
  Week 0 | 5.0 (6.69)
  Week 6: number analyzed (Participants) | 19
  Week 6 | -0.26 (1.759)
  Week 14: number analyzed (Participants) | 17
  Week 14 | -0.35 (2.422)
  Week 26: number analyzed (Participants) | 14
  Week 26 | -0.43 (1.342)

38. Secondary Outcome: Change From Baseline in Short Form (36) Health Survey (SF-36) Domain Average Physical Functioning
Description: Short-form (36) Health Survey domain Average Physical Functioning; scored on a scale of 0-100; lower score equals more disability.
Time Frame: Weeks 0, 2, 6, 10, 14, 18, 22, 26
Population: At baseline (Week 0), the maximum number analyzed was 45. This was the largest N collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 45
score on a scale
  Week 0 | 78.8 (27.92)
  Week 2 | 0.67 (16.011)
  Week 6 | 2.89 (15.576)
  Week 10: number analyzed (Participants) | 43
  Week 10 | 2.09 (16.229)
  Week 14: number analyzed (Participants) | 43
  Week 14 | 5.70 (16.278)
  Week 18: number analyzed (Participants) | 41
  Week 18 | 4.76 (17.028)
  Week 22: number analyzed (Participants) | 37
  Week 22 | 4.05 (15.449)
  Week 26: number analyzed (Participants) | 41
  Week 26 | 4.76 (16.694)

39. Secondary Outcome: Change From Baseline in Short Form (36) Health Survey (SF-36) Domain Average Role Limitations Due to Physical Health
Description: Short-form (36) Health Survey domain Average Role Limitations due to Physical Health; scored on a scale of 0-100; lower score equals more disability.
Time Frame: Weeks 0, 2, 6, 10, 14, 18, 22, 26
Population: At baseline (Week 0), the maximum number analyzed was 45. This was the largest N collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 45
score on a scale
  Week 0 | 72.8 (40.18)
  Week 2 | 0.56 (34.332)
  Week 6 | 11.11 (31.782)
  Week 10: number analyzed (Participants) | 43
  Week 10 | 8.72 (36.954)
  Week 14: number analyzed (Participants) | 43
  Week 14 | 12.21 (36.340)
  Week 18: number analyzed (Participants) | 41
  Week 18 | 10.98 (35.816)
  Week 22: number analyzed (Participants) | 37
  Week 22 | 12.16 (33.136)
  Week 26 | 9.15 (33.427)

40. Secondary Outcome: Change From Baseline in Short Form (36) Health Survey (SF-36) Domain Average Role Limitations Due to Emotional Problems
Description: Short-form (36) Health Survey domain Average Role Limitations due to Emotional Problems; scored on a scale of 0-100; lower score equals more disability.
Time Frame: Weeks 0, 2, 6, 10, 14, 18, 22, 26
Population: At baseline (Week 0), the maximum number analyzed was 45. This was the largest N collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 45
score on a scale
  Week 0 | 76.3 (40.59)
  Week 2 | 7.41 (28.328)
  Week 6 | 9.63 (35.264)
  Week 10: number analyzed (Participants) | 43
  Week 10 | 12.40 (36.387)
  Week 14: number analyzed (Participants) | 43
  Week 14 | 10.85 (36.890)
  Week 18: number analyzed (Participants) | 41
  Week 18 | 11.38 (42.564)
  Week 22: number analyzed (Participants) | 37
  Week 22 | 8.11 (38.814)
  Week 26: number analyzed (Participants) | 41
  Week 26 | 8.13 (36.347)

41. Secondary Outcome: Change From Baseline in Short Form (36) Health Survey (SF-36) Domain Average Energy/Fatigue
Description: Short-form (36) Health Survey domain Average Energy/Fatigue; scored on a scale of 0-100; lower score equals more disability.
Time Frame: Weeks 0, 2, 6, 10, 14, 18, 22, 26
Population: At baseline (Week 0), the maximum number analyzed was 45. This was the largest N collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 45
score on a scale
  Week 0 | 59.7 (26.34)
  Week 2 | 5.44 (19.564)
  Week 6 | 5.89 (16.036)
  Week 10: number analyzed (Participants) | 43
  Week 10 | 9.07 (18.266)
  Week 14: number analyzed (Participants) | 43
  Week 14 | 10.93 (21.220)
  Week 18: number analyzed (Participants) | 41
  Week 18 | 11.59 (22.540)
  Week 22: number analyzed (Participants) | 37
  Week 22 | 9.46 (18.135)
  Week 26: number analyzed (Participants) | 41
  Week 26 | 9.51 (21.148)

42. Secondary Outcome: Change From Baseline in Short Form (36) Health Survey (SF-36) Domain Average Emotional Well-being
Description: Short-form (36) Health Survey domain Average Emotional Well-Being; scored on a scale of 0-100; lower score equals more disability.
Time Frame: Weeks 0, 2, 6, 10, 14, 18, 22, 26
Population: At baseline (Week 0), the maximum number analyzed was 45. This was the largest N collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 45
score on a scale
  Week 0 | 76.4 (16.43)
  Week 2 | 2.93 (14.204)
  Week 6 | 2.84 (12.435)
  Week 10: number analyzed (Participants) | 43
  Week 10 | 6.60 (15.116)
  Week 14: number analyzed (Participants) | 43
  Week 14 | 7.07 (14.757)
  Week 18: number analyzed (Participants) | 41
  Week 18 | 6.24 (17.483)
  Week 22: number analyzed (Participants) | 37
  Week 22 | 5.08 (13.120)
  Week 26: number analyzed (Participants) | 41
  Week 26 | 7.12 (13.342)

43. Secondary Outcome: Change From Baseline in Short Form (36) Health Survey (SF-36) Domain Average Social Functioning
Description: Short-form (36) Health Survey domain Average Social Functioning; scored on a scale of 0-100; lower score equals more disability.
Time Frame: Weeks 0, 2, 6, 10, 14, 18, 22, 26
Population: At baseline (Week 0), the maximum number analyzed was 45. This was the largest N collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 45
score on a scale
  Week 0 | 83.1 (24.01)
  Week 2 | 4.72 (17.935)
  Week 6 | 0.83 (22.519)
  Week 10: number analyzed (Participants) | 43
  Week 10 | 7.85 (21.826)
  Week 14: number analyzed (Participants) | 43
  Week 14 | 5.81 (19.736)
  Week 18: number analyzed (Participants) | 41
  Week 18 | 8.54 (22.611)
  Week 22: number analyzed (Participants) | 37
  Week 22 | 4.73 (16.497)
  Week 26: number analyzed (Participants) | 41
  Week 26 | 5.18 (19.759)

44. Secondary Outcome: Change From Baseline in Short Form (36) Health Survey (SF-36) Domain Average Pain
Description: Short-form (36) Health Survey domain Average Pain; scored on a scale of 0-100; lower score equals more disability.
Time Frame: Weeks 0, 2, 6, 10, 14, 18, 22, 26
Population: At baseline (Week 0), the maximum number analyzed was 45. This was the largest N collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 45
score on a scale
  Week 0 | 74.4 (27.94)
  Week 2 | 6.17 (23.089)
  Week 6 | 6.33 (22.295)
  Week 10: number analyzed (Participants) | 43
  Week 10 | 9.42 (22.729)
  Week 14: number analyzed (Participants) | 43
  Week 14 | 11.57 (19.327)
  Week 18: number analyzed (Participants) | 41
  Week 18 | 9.57 (16.639)
  Week 22: number analyzed (Participants) | 37
  Week 22 | 5.07 (19.225)
  Week 26: number analyzed (Participants) | 41
  Week 26 | 7.80 (18.176)

45. Secondary Outcome: Change From Baseline in Short Form (36) Health Survey (SF-36) Domain Average General Health
Description: Short-form (36) Health Survey domain Average General Health; scored on a scale of 0-100; lower score equals more disability.
Time Frame: Weeks 0, 2, 6, 10, 14, 18, 22, 26
Population: At baseline (Week 0), the maximum number analyzed was 45. This was the largest N collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 45
score on a scale
  Week 0 | 68.2 (27.31)
  Week 2 | 2.44 (15.211)
  Week 6 | 5.00 (17.023)
  Week 10: number analyzed (Participants) | 43
  Week 10 | 6.16 (16.360)
  Week 14: number analyzed (Participants) | 43
  Week 14 | 8.26 (18.577)
  Week 18: number analyzed (Participants) | 41
  Week 18 | 8.05 (19.839)
  Week 22: number analyzed (Participants) | 37
  Week 22 | 6.22 (16.558)
  Week 26: number analyzed (Participants) | 41
  Week 26 | 7.80 (20.002)

46. Secondary Outcome: Change From Baseline in Patient Health Questionnaire 9 (PHQ-9) Total Score
Description: Depression module; scores DSM-IV criteria to monitor severity of depression through 9 total questions; minimum score of 0, maximum score of 27, each question ranges from scores 0-3; higher scores mean worse outcome
Time Frame: Weeks 0, 2, 6, 10, 14, 18, 22, 26
Population: At baseline (Week 0), the maximum number analyzed was 45. This was the largest N collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HB-adMSCs
Number analyzed (Participants) | 45
score on a scale
  Week 0 | 4.9 (6.43)
  Week 2 | -1.67 (5.981)
  Week 6 | -1.24 (5.832)
  Week 10: number analyzed (Participants) | 43
  Week 10 | -2.30 (6.081)
  Week 14: number analyzed (Participants) | 43
  Week 14 | -1.81 (7.433)
  Week 18: number analyzed (Participants) | 41
  Week 18 | -2.68 (5.803)
  Week 22: number analyzed (Participants) | 37
  Week 22 | -2.05 (4.190)
  Week 26: number analyzed (Participants) | 41
  Week 26 | -1.95 (6.569)

ADVERSE EVENTS:
Time Frame: Week 0 (Infusion 1) through Week 26 (End of Study)
Description: 43 out of 51 total subjects experienced at least one adverse event (AE). A total of 154 AEs were recorded during the entirety of the study, 147 of which were mild, 5 moderate, and 2 severe. There were 3 serious adverse events (SAEs) reported during the study period.
Arm/Group | HB-adMSCs
All-Cause Mortality (participants affected / at risk) | 0/51
Serious Adverse Events (participants affected / at risk) | 3/51
Other Adverse Events (participants affected / at risk) | 42/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HB-adMSCs (N=51)
Urinary tract infection (Infections and infestations) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (2)
Embolism (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HB-adMSCs (N=51)
Influenza like illness (General disorders) | 14 (26)
Fatigue (General disorders) | 10 (13)
Pyrexia (General disorders) | 4 (5)
Chills (General disorders) | 2 (5)
Chest pain (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Headache (Nervous system disorders) | 21 (45)
Balance disorder (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Migraine with aura (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Sinus headache (Nervous system disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 (3)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Crohn's disease (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Gastric dilatation (Gastrointestinal disorders) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2)
Herpes zoster (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Palpitations (Cardiac disorders) | 2 (3)
Arrhythmia (Cardiac disorders) | 1 (1)
Vision blurred (Eye disorders) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1)
Blood bicarbonate decreased (Investigations) | 1 (1)
Colonoscopy (Investigations) | 1 (1)
SARS-CoV-2 antibody test positive (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (4)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (3)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-04-20): https://cdn.clinicaltrials.gov/large-docs/31/NCT04349631/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-20): https://cdn.clinicaltrials.gov/large-docs/31/NCT04349631/SAP_001.pdf